CLINICAL TRIAL: NCT00839332
Title: A Phase 1/Randomized Phase 2 Study to Evaluate LY2603618 in Combination With Gemcitabine in Patients With Pancreatic Cancer
Brief Title: A Study for Participants With Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12096; I2I-MC-JMMC (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreas; metastatic cancer; advanced cancer; Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — LY2603618; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2603618 + Gemcitabine (Experimental): Participants participated in Phase 1 or 2.
  LY2603618 (Phase 1): 70 to 250 milligrams/meter squared (mg/m^2) LY2603618 as a 1-hour continuous intravenous (IV) infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until disease progression (DP). Participants received LY2603618 as part of the dose escalation cohort (dose of 70, 105, 150, 200, or 250 mg/m^2) or the expansion cohort (flat dose of 200 mg or 230 mg).
  LY2603618 (Phase 2): 230 mg LY2603618 as a 1-hour continuous IV infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until DP.
  Gemcitabine (Phase 1 and 2): 1000 mg/m^2 gemcitabine as a 30-minute continuous IV infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until DP. Participants received gemcitabine 24 hours prior to LY2603618 administration.
  Interventions: Drug: LY2603618; Drug: Gemcitabine
- Gemcitabine (Active Comparator): Participants participated in Phase 2 only.
  Gemcitabine (Phase 2): 1000 mg/m^2 gemcitabine as a 30-minute continuous IV infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until disease progression.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: LY2603618
  Arms: LY2603618 + Gemcitabine
Drug: Gemcitabine
  Other Names: Gemzar; LY188011

SUMMARY:
The purpose of the Phase 1 portion of this study was to determine the dose of LY2603618 that can be safely administered 24 hours after gemcitabine treatment. This dose was then used for the Phase 2 portion of the study. The Phase 2 portion of the study evaluated whether LY2603618, when administered 24 hours after gemcitabine therapy, was an effective treatment for participants with pancreatic cancer.

DETAILED DESCRIPTION:
Phase 1 included a dose escalation of LY2603618 doses from 70 milligrams/meter squared (mg/m^2) to 250 mg/m^2 divided into 5 cohorts. Each participant was assigned to a single cohort with no intra-participant dose escalation. Phase 1 also included an expansion cohort where participants received a flat dose of 200 or 230 mg LY2603618. Participants received gemcitabine on Days 1, 8, and 15, followed by LY2603618 on Days 2, 9, and 16 of each 28-day cycle. The purpose of the Phase 1 portion was to determine the maximum tolerated LY2603618 dose to be carried into the Phase 2 portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer that is metastatic and/or advanced during Phase 1
* Diagnosed with pancreatic cancer that is metastatic and not amenable to surgery
* Must be at least 18 years of age
* Adequate hematological, liver, and renal functions
* Eastern Cooperative Oncology Group (ECOG) status of 0 to 2

Exclusion Criteria:

* Known hypersensitivity to gemcitabine
* Pregnant or lactating females or refusal to use medically approved contraceptive precautions
* Had prior treatment with radiotherapy involving more than 25% of marrow producing area
* Have received treatment in the last 30 days with a drug which has not received regulatory approval for any indication at the time of study entry

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2009-02; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (30):
- United States (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Macon, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Post Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sioux City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sioux Falls, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tyler, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hampton, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Green Bay, Wisconsin
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heilbronn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nuremberg
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ancona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mendola
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam, Netherlands
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., L'Hospitalet de Llobregat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid

REFERENCES:
- [Derived] Laquente B, Lopez-Martin J, Richards D, Illerhaus G, Chang DZ, Kim G, Stella P, Richel D, Szcylik C, Cascinu S, Frassineti GL, Ciuleanu T, Hurt K, Hynes S, Lin J, Lin AB, Von Hoff D, Calvo E. A phase II study to evaluate LY2603618 in combination with gemcitabine in pancreatic cancer patients. BMC Cancer. 2017 Feb 15;17(1):137. doi: 10.1186/s12885-017-3131-x. PMID 28202004

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: LY2603618 + Gemcitabine: All participants in Phase 1 received LY2603618 in combination with gemcitabine.
  LY2603618: 70 to 250 milligrams/meter squared (mg/m^2) LY2603618 as a 1-hour continuous intravenous (IV) infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until disease progression. Participants received LY2603618 as part of the dose escalation cohort of Phase 1 (dose of 70, 105, 150, 200, or 250 mg/m^2) or as part of the expansion cohort of Phase 1 (flat dose of 200 or 230 mg). The flat dose cohorts were conducted in parallel.
  Gemcitabine: 1000 mg/m^2 gemcitabine as a 30-minute continuous IV infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until disease progression. Participants received gemcitabine 24 hours prior to LY2603618 administration.
- Phase 2: LY2603618 + Gemcitabine: LY2603618: 230 mg flat dose LY2603618 as a 1-hour continuous IV infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until disease progression.
  Gemcitabine: Participants were administered 1000 mg/m^2 gemcitabine as a 30-minute continuous IV infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until disease progression. Participants received gemcitabine 24 hours prior to LY2603618 administration.
- Phase 2: Gemcitabine: Gemcitabine: 1000 mg/m^2 gemcitabine as a 30-minute continuous IV infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until disease progression.
Period: Phase 1
Arm/Group | Phase 1: LY2603618 + Gemcitabine | Phase 2: LY2603618 + Gemcitabine | Phase 2: Gemcitabine
Started | 50 | 0 (Participants in Phase 2 did not participate in Phase 1.) | 0 (Participants in Phase 2 did not participate in Phase 1.)
Received at Least 1 Dose of Study Drug | 50 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 50 | 0 | 0
Not completed — Disease Progression | 38 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: LY2603618 + Gemcitabine | Phase 2: LY2603618 + Gemcitabine | Phase 2: Gemcitabine
Started | 0 (Participants in Phase 1 did not participate in Phase 2.) | 68 | 39
Received at Least 1 Dose of Study Drug | 0 | 65 | 34
Completed | 0 | 0 | 0
Not Completed | 0 | 68 | 39
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Disease Progression | 0 | 46 | 21
Not completed — Adverse Event | 0 | 8 | 6
Not completed — Death | 0 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 5 | 8
Not completed — Physician Decision | 0 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug.
Groups:
- Phase 1: LY2603618 + Gemcitabine: All participants in Phase 1 received LY2603618 in combination with gemcitabine.
  LY2603618: 70 to 250 mg/m^2 LY2603618 as a 1-hour continuous IV infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until disease progression. Participants received LY2603618 as part of the dose escalation cohort of Phase 1 (dose of 70, 105, 150, 200, or 250 mg/m^2) or as part of the expansion cohort of Phase 1 (flat dose of 200 or 230 mg). The flat dose cohorts were conducted in parallel.
  Gemcitabine: 1000 mg/m^2 gemcitabine as a 30-minute continuous IV infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until disease progression. Participants received gemcitabine 24 hours prior to LY2603618 administration.
- Total: Total of all reporting groups
Arm/Group | Phase 1: LY2603618 + Gemcitabine | Phase 2: LY2603618 + Gemcitabine | Phase 2: Gemcitabine | Total
Number analyzed (Participants) | 50 | 65 | 34 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (12.2) | 64.3 (8.3) | 64.4 (10.1) | 62.54 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 14 | 61
  Male | 26 | 42 | 20 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 46 | 62 | 32 | 140
  Black or African American | 1 | 2 | 2 | 5
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 27 | 14 | 73
  Spain | 18 | 12 | 5 | 35
  Romania | 0 | 2 | 1 | 3
  Germany | 0 | 17 | 9 | 26
  Netherlands | 0 | 3 | 2 | 5
  Italy | 0 | 3 | 2 | 5
  Poland | 0 | 1 | 1 | 2
Initial Pathological Diagnosis [Count of Participants; unit: Participants]
  Adenocarcinoma, Pancreas | 10 | 65 | 34 | 109
  Adenocarcinoma, Colon | 7 | 0 | 0 | 7
  Carcinoma, Breast | 4 | 0 | 0 | 4
  Carcinoma, Non-Small Cell, Lung NOS | 3 | 0 | 0 | 3
  Adenocarcinoma, Cervix | 2 | 0 | 0 | 2
  Adenocarcinoma, Rectum | 2 | 0 | 0 | 2
  Carcinoma, Endometrium | 2 | 0 | 0 | 2
  Carcinoma, Infiltrating Ductal, Breast | 2 | 0 | 0 | 2
  Carcinoma, Renal Cell | 2 | 0 | 0 | 2
  Sarcoma, Leiomyosarcoma, Abdomen (Non-Gist) | 2 | 0 | 0 | 2
  Squamous Cell Carcinoma, Head and Neck | 2 | 0 | 0 | 2
  Ampulla of Pancreas | 1 | 0 | 0 | 1
  Carcinoma, Head and Neck | 1 | 0 | 0 | 1
  Carcinoma, Ovarian | 1 | 0 | 0 | 1
  Carcinoma, Peritoneal | 1 | 0 | 0 | 1
  Carcinoma, Small Cell, Lung | 1 | 0 | 0 | 1
  Carcinoma, Transitional Cell, Urothelium | 1 | 0 | 0 | 1
  Ewing's Sarcoma | 1 | 0 | 0 | 1
  Lymphoma, Non-Hodgkin's Lymphoma | 1 | 0 | 0 | 1
  Mesothelioma, Pleural, Malignant | 1 | 0 | 0 | 1
  Ovarian Adenocarcinoma | 1 | 0 | 0 | 1
  Squamous Cell Carcinoma, Cervix | 1 | 0 | 0 | 1
  Tumor | 1 | 0 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death) as follows: 0 - Fully Active; 1 - Ambulatory, Restricted Strenuous Activity; 2 - Ambulatory, No Work Activities; 3 - Partially Confined to Bed, Limited Self Care; 4 - Completely Disabled; and 5 - Dead.
  Participants
    ECOG Status 0 | 19 | 28 | 14 | 61
    ECOG Status 1 | 31 | 31 | 17 | 79
    ECOG Status 2 | 0 | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Determine the Recommended Phase 2 Dose for LY2603618 When Administered After Gemcitabine
Description: The recommended Phase 2 dose for LY2603618 when administered approximately 24 hours after gemcitabine was based on the maximum tolerated dose and achievement of predefined LY2603618 plasma systemic exposures targets (area under the LY2603618 plasma concentration versus time curve from time zero to infinity [AUC(0-inf)] >21,000 nanogram*hour/milliliter [ng*h/mL] and maximum LY2603618 plasma concentration [Cmax] >2000 nanograms/milliliter [ng/mL]).
Time Frame: Baseline through 18 months
Population: Phase 1 participants who received at least 1 dose of study drug.
Measure: Number; unit: milligrams (mg)
Groups:
- Phase 1: LY2603618 + Gemcitabine: All participants in Phase 1 received LY2603618 in combination with gemcitabine.
  LY2603618: 70-250 mg/m^2 LY2603618 as a 1-hour continuous IV infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until disease progression. Participants received LY2603618 as part of the dose escalation cohort of Phase 1 (dose of 70, 105, 150, 200, or 250 mg/m^2) or as part of the expansion cohort of Phase 1 (flat dose of 200 or 230 mg). The flat dose cohorts were conducted in parallel.
  Gemcitabine: 1000 mg/m^2 gemcitabine as a 30-minute continuous IV infusion once per week for 3 weeks, followed by 1 week of rest. This 28-day cycle was repeated for a minimum of 2 cycles and/or until disease progression. Participants received gemcitabine 24 hours prior to LY2603618 administration.
Arm/Group | Phase 1: LY2603618 + Gemcitabine
Number analyzed (Participants) | 50
milligrams (mg) | 230

2. Primary Outcome: Phase 2: Overall Survival (OS)
Description: Overall survival (OS) time is defined as the time from the date of randomization to the date of death from any cause. For participants not known to have died as of the data cut-off date, OS time was censored at the last contact date the participant was known to be alive prior to the cut-off date. OS was summarized using Kaplan-Meier estimates.
Time Frame: Phase 2: Baseline to date of death
Population: Phase 2 participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: LY2603618 + Gemcitabine | Phase 2: Gemcitabine
Number analyzed (Participants) | 65 | 34
months | 7.8 [5.0 to 11.1] | 8.3 [5.1 to 14.1]
Statistical Analysis 1: Comparison: Phase 2: LY2603618 + Gemcitabine vs Phase 2: Gemcitabine; Test type: Superiority or Other; Bayesian Posterior Probability = 0.333 — Inference about survival was made using a Bayesian posterior probability. The combination treatment would have been considered superior to gemcitabine alone if the posterior probability of superiority exceeded 0.8

3. Secondary Outcome: Phase 1: Maximum Plasma Concentration (Cmax) of Gemcitabine, 2',2'-Difluorodeoxyuridine (dFdU), and LY2603618
Description: Plasma samples for pharmacokinetic (PK) analysis were collected following IV infusion of each study drug. However, the dose-normalized PK analysis of gemcitabine and dFdU were not reported because the gemcitabine and dFdU plasma concentration data generated for all participants with PK samples collected in this study were withdrawn (invalidated) as a result of the failure of the Incurred Sample Reanalysis (ISR) for both gemcitabine and dFdU. Therefore, only the LY2603618 plasma Cmax values are reported for each LY2603618 dose level on Cycle (C) 1 /Day (D) 1, Cycle 1 /Day 16, and Cycle 2 /Day 2. The number of PK observations (n) used in the analysis is presented for each dose level and time point.
Time Frame: Phase 1: LY2603618 - Predose and 0, 1, 3, 6, 24, 48, and 72 hours after the end of infusion on C1 /D2, C1 /D16, and C2 /D2. Gemcitabine - Predose and 0, 10, 30, 60, and 120 minutes after the end of infusion on C1 /D1, C1 /D15, and C2 /D1.
Population: Phase 1 participants who received at least 1 dose of study drug (LY2603618) and had sufficient LY2603618 plasma concentration data to enable determination of the LY2603618 Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Phase 1: LY2603618 + Gemcitabine
Number analyzed (Participants) | 50
nanograms per milliliter (ng/mL)
  70 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 2
  70 mg/m^2, Cycle 1 /Day 2 | 3530 (23)
  70 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 3
  70 mg/m^2, Cycle 1 /Day 16 | 3360 (26)
  70 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 3
  70 mg/m^2, Cycle 2 /Day 2 | 3100 (12)
  105 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 3
  105 mg/m^2, Cycle 1 /Day 2 | 4890 (25)
  105 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 3
  105 mg/m^2, Cycle 1 /Day 16 | 5170 (38)
  105 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 3
  105 mg/m^2, Cycle 2 /Day 2 | 5360 (23)
  150 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 7
  150 mg/m^2, Cycle 1 /Day 2 | 4280 (29)
  150 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 6
  150 mg/m^2, Cycle 1 /Day 16 | 5040 (38)
  150 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 6
  150 mg/m^2, Cycle 2 /Day 2 | 4370 (38)
  200 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 11
  200 mg/m^2, Cycle 1 /Day 2 | 4870 (63)
  200 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 8
  200 mg/m^2, Cycle 1 /Day 16 | 5360 (40)
  200 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 11
  200 mg/m^2, Cycle 2 /Day 2 | 5290 (40)
  250 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 5
  250 mg/m^2, Cycle 1 /Day 2 | 7990 (25)
  250 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 3
  250 mg/m^2, Cycle 1 /Day 16 | 7990 (6)
  250 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 3
  250 mg/m^2, Cycle 2 /Day 2 | 5290 (35)
  200 mg (flat dose), Cycle 1 /Day 2: number analyzed (Participants) | 10
  200 mg (flat dose), Cycle 1 /Day 2 | 3440 (65)
  200 mg (flat dose), Cycle 1 /Day 16: number analyzed (Participants) | 6
  200 mg (flat dose), Cycle 1 /Day 16 | 3470 (61)
  200 mg (flat dose), Cycle 2 /Day 2: number analyzed (Participants) | 8
  200 mg (flat dose), Cycle 2 /Day 2 | 3640 (45)
  230 mg (flat dose), Cycle 1 /Day 2: number analyzed (Participants) | 10
  230 mg (flat dose), Cycle 1 /Day 2 | 4820 (72)
  230 mg (flat dose), Cycle 1 /Day 16: number analyzed (Participants) | 6
  230 mg (flat dose), Cycle 1 /Day 16 | 4980 (35)
  230 mg (flat dose), Cycle 2 /Day 2: number analyzed (Participants) | 7
  230 mg (flat dose), Cycle 2 /Day 2 | 3830 (26)

4. Secondary Outcome: Phase 2: Maximum Plasma Concentration (Cmax) of Gemcitabine, dFdU, and LY2603618
Description: Plasma samples for PK analysis were collected following IV infusion of each study drug. However, the dose-normalized PK analysis of gemcitabine and dFdU were not reported because the gemcitabine and dFdU plasma concentration data generated for all participants with PK samples collected in this study were withdrawn (invalidated) as a result of the failure of the Incurred Sample Reanalysis (ISR) for both gemcitabine and dFdU. Therefore, only the LY2603618 plasma Cmax values are reported at the 230 mg LY2603618 dose level on Cycle 1 /Day 1, Cycle 1 /Day 16, and Cycle 2 /Day 2. The number of PK observations (n) used in the analysis is presented for each time point.
Time Frame: Phase 2: LY2603618 - Predose and 0, 1, 3, and 24 hours after the end of infusion on Days 2 and 16 of Cycle 1. Gemcitabine - Predose and 0, 10, 60, and 120 minutes after the end of infusion on Days 1 and 15 of Cycle 1.
Population: Phase 2 participants who received at least 1 dose of study drug (LY2603618) and had sufficient LY2603618 plasma concentration data to enable determination of the LY2603618 Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 2: LY2603618 + Gemcitabine
Number analyzed (Participants) | 62
ng/mL
  Cycle 1 /Day 2: number analyzed (Participants) | 58
  Cycle 1 /Day 2 | 3170 (50)
  Cycle 1 /Day 16: number analyzed (Participants) | 48
  Cycle 1 /Day 16 | 3410 (50)
  Cycle 2 /Day 2: number analyzed (Participants) | 2
  Cycle 2 /Day 2 | 2390 (54)

5. Secondary Outcome: Phase 1: Area Under the Plasma Concentration Versus Time Curve (AUC) of Gemcitabine, dFdU, and LY2603618
Description: Plasma samples for PK analysis were collected following IV infusion of each study drug. However, the dose-normalized PK analysis of gemcitabine and dFdU were not reported because the gemcitabine plasma and dFdU concentration data generated for all participants with PK samples collected in this study were withdrawn (invalidated) as a result of the failure of the Incurred Sample Reanalysis (ISR) for both gemcitabine and dFdU. Therefore, only LY2603618 plasma AUC from time zero to 24 hours (AUC[0-24]), AUC from time zero to the last time point with a measurable concentration (AUC[0-tlast]), and AUC from time zero to infinity (AUC[0-inf]) values are reported for each LY2603618 dose level on Cycle 1 /Day 1, Cycle 1 /Day 16, and Cycle 2 /Day 2. The number of PK observations (n) used in the analysis is presented for each dose level and time point.
Time Frame: as for outcome 3
Population: Phase 1 participants who received at least 1 dose of study drug (LY2603618) and had sufficient LY2603618 plasma concentration data to enable calculation of the LY2603618 AUC.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Arm/Group | Phase 1: LY2603618 + Gemcitabine
Number analyzed (Participants) | 50
nanogram*hour/milliliter (ng*h/mL)
  AUC(0-24), 70 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 2
  AUC(0-24), 70 mg/m^2, Cycle 1 /Day 2 | 21300 (24)
  AUC(0-24), 70 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 3
  AUC(0-24), 70 mg/m^2, Cycle 1 /Day 16 | 21200 (27)
  AUC(0-24), 70 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 3
  AUC(0-24), 70 mg/m^2, Cycle 2 /Day 2 | 19900 (24)
  AUC(0-24), 105 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 3
  AUC(0-24), 105 mg/m^2, Cycle 1 /Day 2 | 40500 (23)
  AUC(0-24), 105 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 3
  AUC(0-24), 105 mg/m^2, Cycle 1 /Day 16 | 50100 (32)
  AUC(0-24), 105 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 3
  AUC(0-24), 105 mg/m^2, Cycle 2 /Day 2 | 49800 (4)
  AUC(0-24), 150 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 7
  AUC(0-24), 150 mg/m^2, Cycle 1 /Day 2 | 32200 (27)
  AUC(0-24), 150 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 6
  AUC(0-24), 150 mg/m^2, Cycle 1 /Day 16 | 40000 (29)
  AUC(0-24), 150 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 6
  AUC(0-24), 150 mg/m^2, Cycle 2 /Day 2 | 31000 (42)
  AUC(0-24), 200 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 10
  AUC(0-24), 200 mg/m^2, Cycle 1 /Day 2 | 40200 (42)
  AUC(0-24), 200 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 8
  AUC(0-24), 200 mg/m^2, Cycle 1 /Day 16 | 39800 (36)
  AUC(0-24), 200 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 11
  AUC(0-24), 200 mg/m^2, Cycle 2 /Day 2 | 44300 (39)
  AUC(0-24), 250 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 5
  AUC(0-24), 250 mg/m^2, Cycle 1 /Day 2 | 88800 (27)
  AUC(0-24), 250 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 3
  AUC(0-24), 250 mg/m^2, Cycle 1 /Day 16 | 61000 (63)
  AUC(0-24), 250 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 3
  AUC(0-24), 250 mg/m^2, Cycle 2 /Day 2 | 40000 (112)
  AUC(0-24), 200 mg (flat), Cycle 1 /Day 2: number analyzed (Participants) | 10
  AUC(0-24), 200 mg (flat), Cycle 1 /Day 2 | 22900 (77)
  AUC(0-24), 200 mg (flat), Cycle 1 /Day 16: number analyzed (Participants) | 6
  AUC(0-24), 200 mg (flat), Cycle 1 /Day 16 | 28700 (63)
  AUC(0-24), 200 mg (flat), Cycle 2 /Day 2: number analyzed (Participants) | 8
  AUC(0-24), 200 mg (flat), Cycle 2 /Day 2 | 23800 (62)
  AUC(0-24), 230 mg (flat), Cycle 1 /Day 2: number analyzed (Participants) | 10
  AUC(0-24), 230 mg (flat), Cycle 1 /Day 2 | 32400 (38)
  AUC(0-24), 230 mg (flat), Cycle 1 /Day 16: number analyzed (Participants) | 6
  AUC(0-24), 230 mg (flat), Cycle 1 /Day 16 | 32300 (22)
  AUC(0-24), 230 mg (flat), Cycle 2 /Day 2: number analyzed (Participants) | 7
  AUC(0-24), 230 mg (flat), Cycle 2 /Day 2 | 32500 (24)
  AUC(0-tlast), 70 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 2
  AUC(0-tlast), 70 mg/m^2, Cycle 1 /Day 2 | 24600 (28)
  AUC(0-tlast), 70 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 3
  AUC(0-tlast), 70 mg/m^2, Cycle 1 /Day 16 | 27500 (21)
  AUC(0-tlast), 70 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 3
  AUC(0-tlast), 70 mg/m^2, Cycle 2 /Day 2 | 25800 (29)
  AUC(0-tlast), 105 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 3
  AUC(0-tlast), 105 mg/m^2, Cycle 1 /Day 2 | 65800 (53)
  AUC(0-tlast), 105 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 3
  AUC(0-tlast), 105 mg/m^2, Cycle 1 /Day 16 | 75500 (46)
  AUC(0-tlast), 105 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 3
  AUC(0-tlast), 105 mg/m^2, Cycle 2 /Day 2 | 79600 (19)
  AUC(0-tlast), 150 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 7
  AUC(0-tlast), 150 mg/m^2, Cycle 1 /Day 2 | 41600 (31)
  AUC(0-tlast), 150 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 6
  AUC(0-tlast), 150 mg/m^2, Cycle 1 /Day 16 | 52000 (38)
  AUC(0-tlast), 150 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 6
  AUC(0-tlast), 150 mg/m^2, Cycle 2 /Day 2 | 39800 (45)
  AUC(0-tlast), 200 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 11
  AUC(0-tlast), 200 mg/m^2, Cycle 1 /Day 2 | 44300 (85)
  AUC(0-tlast), 200 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 8
  AUC(0-tlast), 200 mg/m^2, Cycle 1 /Day 16 | 55300 (51)
  AUC(0-tlast), 200 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 11
  AUC(0-tlast), 200 mg/m^2, Cycle 2 /Day 2 | 55600 (51)
  AUC(0-tlast), 250 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 5
  AUC(0-tlast), 250 mg/m^2, Cycle 1 /Day 2 | 140000 (37)
  AUC(0-tlast), 250 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 3
  AUC(0-tlast), 250 mg/m^2, Cycle 1 /Day 16 | 98200 (139)
  AUC(0-tlast), 250 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 3
  AUC(0-tlast), 250 mg/m^2, Cycle 2 /Day 2 | 60400 (178)
  AUC(0-tlast), 200 mg (flat), Cycle 1 /Day 2: number analyzed (Participants) | 10
  AUC(0-tlast), 200 mg (flat), Cycle 1 /Day 2 | 33100 (101)
  AUC(0-tlast), 200 mg (flat), Cycle 1 /Day 16: number analyzed (Participants) | 6
  AUC(0-tlast), 200 mg (flat), Cycle 1 /Day 16 | 42600 (88)
  AUC(0-tlast), 200 mg (flat), Cycle 2 /Day 2: number analyzed (Participants) | 8
  AUC(0-tlast), 200 mg (flat), Cycle 2 /Day 2 | 32400 (85)
  AUC(0-tlast), 230 mg (flat), Cycle 1 /Day 2: number analyzed (Participants) | 10
  AUC(0-tlast), 230 mg (flat), Cycle 1 /Day 2 | 43000 (50)
  AUC(0-tlast), 230 mg (flat), Cycle 1 /Day 16: number analyzed (Participants) | 6
  AUC(0-tlast), 230 mg (flat), Cycle 1 /Day 16 | 51900 (50)
  AUC(0-tlast), 230 mg (flat), Cycle 2 /Day 2: number analyzed (Participants) | 7
  AUC(0-tlast), 230 mg (flat), Cycle 2 /Day 2 | 45900 (26)
  AUC(0-inf), 70 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 2
  AUC(0-inf), 70 mg/m^2, Cycle 1 /Day 2 | 24900 (29)
  AUC(0-inf), 70 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 3
  AUC(0-inf), 70 mg/m^2, Cycle 1 /Day 16 | 28600 (19)
  AUC(0-inf), 70 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 3
  AUC(0-inf), 70 mg/m^2, Cycle 2 /Day 2 | 27100 (31)
  AUC(0-inf), 105 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 3
  AUC(0-inf), 105 mg/m^2, Cycle 1 /Day 2 | 78600 (68)
  AUC(0-inf), 105 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 3
  AUC(0-inf), 105 mg/m^2, Cycle 1 /Day 16 | 79800 (51)
  AUC(0-inf), 105 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 3
  AUC(0-inf), 105 mg/m^2, Cycle 2 /Day 2 | 88800 (25)
  AUC(0-inf), 150 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 7
  AUC(0-inf), 150 mg/m^2, Cycle 1 /Day 2 | 42800 (33)
  AUC(0-inf), 150 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 6
  AUC(0-inf), 150 mg/m^2, Cycle 1 /Day 16 | 54600 (43)
  AUC(0-inf), 150 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 6
  AUC(0-inf), 150 mg/m^2, Cycle 2 /Day 2 | 41000 (46)
  AUC(0-inf), 200 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 10
  AUC(0-inf), 200 mg/m^2, Cycle 1 /Day 2 | 60300 (58)
  AUC(0-inf), 200 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 8
  AUC(0-inf), 200 mg/m^2, Cycle 1 /Day 16 | 56800 (54)
  AUC(0-inf), 200 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 11
  AUC(0-inf), 200 mg/m^2, Cycle 2 /Day 2 | 65400 (49)
  AUC(0-inf), 250 mg/m^2, Cycle 1 /Day 2: number analyzed (Participants) | 5
  AUC(0-inf), 250 mg/m^2, Cycle 1 /Day 2 | 153000 (41)
  AUC(0-inf), 250 mg/m^2, Cycle 1 /Day 16: number analyzed (Participants) | 3
  AUC(0-inf), 250 mg/m^2, Cycle 1 /Day 16 | 101000 (141)
  AUC(0-inf), 250 mg/m^2, Cycle 2 /Day 2: number analyzed (Participants) | 3
  AUC(0-inf), 250 mg/m^2, Cycle 2 /Day 2 | 70500 (216)
  AUC(0-inf), 200 mg (flat), Cycle 1 /Day 2: number analyzed (Participants) | 10
  AUC(0-inf), 200 mg (flat), Cycle 1 /Day 2 | 35200 (117)
  AUC(0-inf), 200 mg (flat), Cycle 1 /Day 16: number analyzed (Participants) | 6
  AUC(0-inf), 200 mg (flat), Cycle 1 /Day 16 | 45700 (93)
  AUC(0-inf), 200 mg (flat), Cycle 2 /Day 2: number analyzed (Participants) | 8
  AUC(0-inf), 200 mg (flat), Cycle 2 /Day 2 | 34400 (93)
  AUC(0-inf), 230 mg (flat), Cycle 1 /Day 2: number analyzed (Participants) | 10
  AUC(0-inf), 230 mg (flat), Cycle 1 /Day 2 | 45200 (50)
  AUC(0-inf), 230 mg (flat), Cycle 1 /Day 16: number analyzed (Participants) | 6
  AUC(0-inf), 230 mg (flat), Cycle 1 /Day 16 | 57700 (58)
  AUC(0-inf), 230 mg (flat), Cycle 2 /Day 2: number analyzed (Participants) | 7
  AUC(0-inf), 230 mg (flat), Cycle 2 /Day 2 | 48000 (26)

6. Secondary Outcome: Phase 2: Area Under the Plasma Concentration Versus Time Curve (AUC) of Gemcitabine, dFdU, and LY2603618
Description: Plasma samples for PK analysis were collected following IV infusion of each study drug. However, the dose-normalized PK analysis of gemcitabine and dFdU were not reported because the gemcitabine and dFdU plasma concentration data generated for all participants with PK samples collected in this study were withdrawn (invalidated) as a result of the failure of the Incurred Sample Reanalysis (ISR) for both gemcitabine and dFdU. Therefore, only the LY2603618 plasma AUC(0-24), AUC(0-tlast), and AUC(0-inf) values are reported for the 230 mg LY2603618 dose on Cycle 1 /Day 1, Cycle 1 /Day 16, and Cycle 2 /Day 2. The number of PK observations (n) used in the analysis is presented for each time point.
Time Frame: as for outcome 4
Population: Phase 2 participants who received at least 1 dose of study drug (LY2603618) and had sufficient LY2603618 plasma concentration data to enable calculation of the LY2603618 AUC.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 2: LY2603618 + Gemcitabine
Number analyzed (Participants) | 62
ng*h/mL
  AUC(0-24), Cycle 1 /Day 2: number analyzed (Participants) | 54
  AUC(0-24), Cycle 1 /Day 2 | 23200 (68)
  AUC(0-24), Cycle 1 /Day 16: number analyzed (Participants) | 42
  AUC(0-24), Cycle 1 /Day 16 | 23700 (60)
  AUC(0-24), Cycle 2 /Day 2: number analyzed (Participants) | 2
  AUC(0-24), Cycle 2 /Day 2 | 19800 (63)
  AUC(0-tlast), Cycle 1 /Day 2: number analyzed (Participants) | 58
  AUC(0-tlast), Cycle 1 /Day 2 | 22200 (73)
  AUC(0-tlast), Cycle 1 /Day 16: number analyzed (Participants) | 48
  AUC(0-tlast), Cycle 1 /Day 16 | 20800 (78)
  AUC(0-tlast), Cycle 2 /Day 2: number analyzed (Participants) | 2
  AUC(0-tlast), Cycle 2 /Day 2 | 20100 (64)
  AUC(0-inf), Cycle 1 /Day 2: number analyzed (Participants) | 54
  AUC(0-inf), Cycle 1 /Day 2 | 29400 (84)
  AUC(0-inf), Cycle 1 /Day 16: number analyzed (Participants) | 42
  AUC(0-inf), Cycle 1 /Day 16 | 29100 (74)
  AUC(0-inf), Cycle 2 /Day 2: number analyzed (Participants) | 2
  AUC(0-inf), Cycle 2 /Day 2 | 23300 (69)

7. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) time was defined as the time from the date of randomization to the first date of progressive disease (symptomatic or objective) or death due to any cause, whichever occurred first. For participants who were not known to have died or progressed as of the data-inclusion cutoff date, PFS time was censored at the date of the last objective progression-free disease assessment prior to the date of any subsequent systematic anticancer therapy. PFS was summarized using Kaplan-Meier estimates.
Time Frame: Phase 2: Baseline to measured progressive disease or date of death from any cause
Population: Phase 2 participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: LY2603618 + Gemcitabine | Phase 2: Gemcitabine
Number analyzed (Participants) | 65 | 34
months | 3.5 [2.1 to 3.6] | 5.6 [2.6 to 7.6]

8. Secondary Outcome: Phase 2: Overall Response Rate
Description: Overall response rate is the best response of complete response (CR) or partial response (PR) as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1) guidelines. CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of not-target lesions or appearance of new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: Phase 2: Baseline to measured progressive disease or date of death from any cause
Population: Phase 2 participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: LY2603618 + Gemcitabine | Phase 2: Gemcitabine
Number analyzed (Participants) | 65 | 34
percentage of participants | 21.5 [12.3 to 33.5] | 8.8 [1.9 to 23.7]

9. Secondary Outcome: Phase 2: Clinical Benefit Rate
Description: Clinical benefit rate is the best response CR, PR, or stable disease (SD) as classified by the investigators according to the RECIST v1.1 guidelines. CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of not-target lesions or appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameter since treatment started. Overall response rate is calculated as a total number of participants with CR, PR, or SD divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: Phase 2: Baseline to measured progressive disease or date of death from any cause
Population: Phase 2 participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: LY2603618 + Gemcitabine | Phase 2: Gemcitabine
Number analyzed (Participants) | 65 | 34
percentage of participants | 55.4 [42.5 to 67.7] | 64.7 [46.5 to 80.3]

10. Other Pre Specified Outcome: Number of Deaths During the Phase 1 Post-study Period
Description: The number of participants who died during the post-study period of Phase 1 does not include the outcomes for the 4 participants who died while on treatment during Phase 2 as captured in the Participant Flow Table. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Phase 1: Time of last dose of study drug through the end of the follow-up period
Population: Participants enrolled in Phase 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: LY2603618 + Gemcitabine
Number analyzed (Participants) | 50
Participants
  Total deaths | 5
  Deaths within 30 days of last dose of study drug | 4
  Deaths during the follow-up period | 1

11. Secondary Outcome: Phase 2: Duration of Response
Description: Duration of response was defined as the time from the first observation of complete response (CR) or partial response (PR) to the first observation of progressive disease or death from any cause. For participants who were not known to have died as of the data-inclusion cut-off date and who do not have progressive disease, the duration was censored at the date of the last objective progression-free disease assessment prior to the date of any subsequent anticancer therapy (systemic, radiologic, or surgery). Participants were also censored at the last valid assessment prior to missing more than 1 consecutive scheduled assessment. Duration of response was summarized using Kaplan-Meier estimates.
Time Frame: Phase 2. Baseline to measured progressive disease or date of death from any cause
Population: Phase 2 participants who received at least 1 dose of study drug and had a confirmed response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: LY2603618 + Gemcitabine | Phase 2: Gemcitabine
Number analyzed (Participants) | 14 | 3
months | 3.5 [1.9 to 5.8] | 6.0 [3.7 to 6.8]

12. Secondary Outcome: Phase 1: Electrocardiogram QTc Prolongation
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave. Twelve-lead electrocardiogram (ECG) data was used to calculate the corrected QT (QTc) based on Fridericia's formula (QTc=QT/RR^0.33, where RR is the interval between two R waves). For each participant, changes in QTc were calculated by subtracting the reading taken before LY2603618 administration from the reading taken after LY2603618 administration on Days 2 and 16 during Cycle 1. The number of participants in which the change in QTc was <=30 milliseconds (msec), >30-60 msec, or >60 msec is presented by dose group and overall.
Time Frame: Phase 1: Days 2 and 16 of Cycle 1
Population: Phase 1 participants who received at least 1 dose of LY2603618 and had evaluable ECG data.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: LY2603618 + Gemcitabine
Number analyzed (Participants) | 49
Participants
  70 mg/m^2, <=30 msec: number analyzed (Participants) | 3
  70 mg/m^2, <=30 msec | 2
  70 mg/m^2, >30-60 msec: number analyzed (Participants) | 3
  70 mg/m^2, >30-60 msec | 1
  70 mg/m^2, >60 msec: number analyzed (Participants) | 3
  70 mg/m^2, >60 msec | 0
  105 mg/m^2, <=30 msec: number analyzed (Participants) | 3
  105 mg/m^2, <=30 msec | 2
  105 mg/m^2, >30-60 msec: number analyzed (Participants) | 3
  105 mg/m^2, >30-60 msec | 0
  105 mg/m^2, >60 msec: number analyzed (Participants) | 3
  105 mg/m^2, >60 msec | 0
  150 mg/m^2, <=30 msec: number analyzed (Participants) | 7
  150 mg/m^2, <=30 msec | 6
  150 mg/m^2, >30-60 msec: number analyzed (Participants) | 7
  150 mg/m^2, >30-60 msec | 1
  150 mg/m^2, >60 msec: number analyzed (Participants) | 7
  150 mg/m^2, >60 msec | 0
  200 mg/m^2, <=30 msec: number analyzed (Participants) | 11
  200 mg/m^2, <=30 msec | 11
  200 mg/m^2, >30-60 msec: number analyzed (Participants) | 11
  200 mg/m^2, >30-60 msec | 0
  200 mg/m^2, >60 msec: number analyzed (Participants) | 11
  200 mg/m^2, >60 msec | 0
  250 mg/m^2, <=30 msec: number analyzed (Participants) | 6
  250 mg/m^2, <=30 msec | 6
  250 mg/m^2, >30-60 msec: number analyzed (Participants) | 6
  250 mg/m^2, >30-60 msec | 0
  250 mg/m^2, >60 msec: number analyzed (Participants) | 6
  250 mg/m^2, >60 msec | 0
  200 mg (flat dose), <=30 msec: number analyzed (Participants) | 10
  200 mg (flat dose), <=30 msec | 9
  200 mg (flat dose), >30-60 msec: number analyzed (Participants) | 10
  200 mg (flat dose), >30-60 msec | 1
  200 mg (flat dose), >60 msec: number analyzed (Participants) | 10
  200 mg (flat dose), >60 msec | 0
  230 mg (flat dose), <=30 msec: number analyzed (Participants) | 10
  230 mg (flat dose), <=30 msec | 8
  230 mg (flat dose), >30-60 msec: number analyzed (Participants) | 10
  230 mg (flat dose), >30-60 msec | 2
  230 mg (flat dose), >60 msec: number analyzed (Participants) | 10
  230 mg (flat dose), >60 msec | 0
  Total, <=30 msec | 44
  Total, >30-60 msec | 5
  Total, >60 msec | 0

13. Secondary Outcome: Phase 2: Electrocardiogram QTc Prolongation
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave. Twelve-lead ECG data was used to calculate QTc based on Fridericia's formula (QTc=QT/RR^0.33, where RR is the interval between two R waves). For each participant, changes in QTc were calculated by subtracting the reading taken before LY2603618 administration from the reading taken after LY2603618 administration on Days 2 and 16 during Cycle 1. The number of participants in which the change in QTc was <=30 milliseconds (msec), >30-60 msec, or >60 msec is presented.
Time Frame: Phase 2: Days 2 and 16 of Cycle 1
Population: Phase 2 participants who received at least 1 dose of LY2603618 and had evaluable ECG data.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: LY2603618 + Gemcitabine
Number analyzed (Participants) | 60
Participants
  <=30 msec | 55
  >30-60 msec | 5
  >60 msec | 0

ADVERSE EVENTS:
Arm/Group | Phase 1: LY2603618 + Gemcitabine | Phase 2: LY2603618 + Gemcitabine | Phase 2: Gemcitabine
Serious Adverse Events (participants affected / at risk) | 21/50 | 27/65 | 18/34
Other Adverse Events (participants affected / at risk) | 48/50 | 64/65 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 1: LY2603618 + Gemcitabine (N=50) | Phase 2: LY2603618 + Gemcitabine (N=65) | Phase 2: Gemcitabine (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (2)
Device occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 2 (2)
Thrombosis in device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 3 (3) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/24 (0) | 0/23 (0) | 1/14 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Phlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: LY2603618 + Gemcitabine (N=50) | Phase 2: LY2603618 + Gemcitabine (N=65) | Phase 2: Gemcitabine (N=34)
Anaemia (Blood and lymphatic system disorders) | 23 (29) | 16 (21) | 10 (13)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 4 (5) | 8 (27) | 6 (10)
Lymphopenia (Blood and lymphatic system disorders) | 5 (6) | 4 (7) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 16 (26) | 15 (49) | 10 (24)
Thrombocytopenia (Blood and lymphatic system disorders) | 23 (46) | 23 (63) | 15 (39)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (5)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 2 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 12 (12) | 14 (19) | 5 (7)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 17 (22) | 21 (27) | 9 (10)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 21 (36) | 10 (15)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 4 (7) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 20 (25) | 27 (42) | 15 (21)
Steatorrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 5 (9) | 13 (14) | 2 (2)
Vomiting (Gastrointestinal disorders) | 14 (16) | 19 (35) | 4 (5)
Asthenia (General disorders) | 4 (5) | 10 (19) | 5 (8)
Chills (General disorders) | 5 (6) | 9 (15) | 2 (2)
Fatigue (General disorders) | 31 (50) | 22 (28) | 14 (19)
Influenza like illness (General disorders) | 3 (3) | 3 (8) | 3 (3)
Infusion site pain (General disorders) | 5 (10) | 0 (0) | 1 (4)
Irritability (General disorders) | 3 (3) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 8 (9) | 19 (23) | 12 (16)
Pyrexia (General disorders) | 15 (33) | 19 (23) | 11 (14)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 2 (2) | 4 (4)
Drug hypersensitivity (Immune system disorders) | 5 (5) | 2 (5) | 0 (0)
Oral candidiasis (Infections and infestations) | 4 (4) | 1 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 10 (15) | 13 (18) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 11 (14) | 10 (15) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 5 (5) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 12 (12) | 3 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 2 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (3) | 2 (6)
Platelet count decreased (Investigations) | 0 (0) | 7 (11) | 1 (5)
Weight decreased (Investigations) | 2 (3) | 7 (8) | 3 (3)
White blood cell count decreased (Investigations) | 2 (2) | 2 (4) | 2 (8)
Decreased appetite (Metabolism and nutrition disorders) | 16 (19) | 21 (22) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (8) | 12 (13) | 4 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 4 (4) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 5 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 6 (7) | 5 (5)
Hypovolaemia (Metabolism and nutrition disorders) | 4 (8) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (10) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 (9) | 2 (2) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7) | 8 (9) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 5 (5) | 5 (5) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (5) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 5 (7) | 7 (10) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 7 (8) | 2 (4)
Anxiety (Psychiatric disorders) | 4 (4) | 0 (0) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 6 (7) | 2 (2) | 3 (4)
Insomnia (Psychiatric disorders) | 7 (9) | 4 (4) | 6 (8)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 7 (7) | 5 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 12 (13) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (8) | 5 (6)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (6) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 4 (4) | 3 (3)
Flushing (Vascular disorders) | 6 (8) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 3 (3)
Hypotension (Vascular disorders) | 5 (5) | 3 (3) | 5 (5)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days